CLINICAL TRIAL: NCT00676663
Title: A Phase 2, Randomized, Double-Blind, Multicenter Study of Exemestane With and Without SNDX-275 in Postmenopausal Women With Locally Recurrent or Metastatic Estrogen Receptor-Positive Breast Cancer, Progressing on Treatment With a Non-Steroidal Aromatase Inhibitor
Brief Title: Study to Evaluate Exemestane With and Without Entinostat (SNDX-275) in Treatment of Postmenopausal Women With Advanced Breast Cancer
Acronym: ENCORE301
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNDX-275-0301; 2009-012623-28 (EudraCT Number)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer; Estrogen Receptor-Positive Breast Cancer; Breast Cancer, Estrogen Receptor-Positive; ER+ Breast Cancer
Keywords: Breast Neoplasms; Breast Tumor; Mammary Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Mammary Neoplasms, Animal | interventions — entinostat; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exemestane 25 mg + Entinostat 5 mg (Experimental): Exemestane (Aromasin®) 25 mg tablets orally once daily plus an entinostat 5 mg tablet orally once per week on Days 1, 8, 15 and 22 of each 28-day treatment cycle until development of progressive disease (PD) or unacceptable toxicity or closure of the study by the Sponsor, whichever occurred first.
  Interventions: Drug: entinostat; Drug: exemestane
- Exemestane 25 mg + Placebo (Placebo Comparator): Exemestane (Aromasin®) 25 mg tablets orally once daily plus a placebo-matching entinostat tablet orally once per week on Days 1, 8, 15 and 22 of each 28-day treatment cycle until development of progressive disease (PD) or unacceptable toxicity or closure of the study by the Sponsor, whichever occurred first.
  Interventions: Drug: exemestane; Drug: Placebo

INTERVENTIONS:
Drug: entinostat — Entinostat 5 mg tablet orally once per week
  Other Names: SNDX-275
  Arms: Exemestane 25 mg + Entinostat 5 mg
Drug: exemestane — Exemestane 25 mg tablet orally once daily
  Other Names: Aromasin®
Drug: Placebo — Placebo-matching entinostat tablet orally once per week
  Arms: Exemestane 25 mg + Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of entinostat in combination with exemestane in the treatment of advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female patients
* Histologically or cytologically confirmed estrogen receptor positive (ER+) breast cancer
* Relapsed or progressed on prior treatment with aromatase inhibitor (AI)
* Metastatic disease must be measurable
* Patients receiving palliative radiation at the non-target lesions must have a 2 week wash out period following completion of the treatment prior to enrollment
* Patient may have had one prior chemotherapy as part of first line therapy as long as it was received before initiation of prior AI
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 1
* Laboratory parameters: a)Hemoglobin ≥ 9.0 g/dL; platelets ≥ 100.0 x 10^9/L; Absolute Neutrophil Count (ANC ≥) 1.5 x 10^9/L without the use of hematopoietic growth factors b)Creatinine less than 2.5 times the upper limit of normal for the institution c)Aspartate transaminase (AST) and alanine transaminase (ALT) less than 2.5 times the upper limit of normal for the institution
* Able to understand and give written informed consent and comply with study procedures

Exclusion Criteria:

* Relapse on treatment with non-steroidal AI after less than 12 months for patients in the adjuvant setting
* Progressive disease after less than 3 months treatment with most recent AI for patients with metastatic disease
* Rapidly progressive, life-threatening metastases
* Any palliative radiotherapy to the measurable lesion
* Previous treatment with SNDX-275 or any other histone deacetylase (HDAC) inhibitor including valproic acid
* Allergy to benzamides or inactive components of the study drug
* A history of allergies to any active or inactive ingredients of exemestane
* Any concomitant medical condition that precludes adequate study treatment compliance
* Patient is currently enrolled in (or completed within 30 days before study drug administration) another investigational drug study
* Patient is currently receiving treatment with valproic acid, Zolinza (vorinostat) or any other HDAC inhibitor or deoxyribonucleic acid (DNA) methyltransferase inhibitor or any systemic anticancer treatment (with the exception of Lupron)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-06-13 (Actual); Primary Completion 2011-01-29 (Actual); Study Completion 2012-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Yardley, MD, Principal Investigator — Sarah Cannon Cancer Center
Locations (38):
- United States (24):
  - California Cancer Care, Greenbrae, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Scripps Health, La Jolla, California
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - University of Southern Florida -Moffitt Cancer Center, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Indiana University Indiana Cancer Pavilion, Indianapolis, Indiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Kansas City Cancer Center, Kansas City, Missouri
  - Hematology-Oncology Associates of Northern New Jersey, Morristown, New Jersey
  - Carolinas Healthcare System Clinical Trials, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - South Texas Cancer Center, McAllen, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Columbia Basin Hematology & Oncology, Kennewick, Washington
  - Puget Sound Cancer Center, Seattle, Washington
- Canada (2):
  - RSM Durham Regional Cancer Center - Lakeridge Health, Oshawa, Ontario
  - St. Joseph's Health Centre, Toronto, Ontario
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Radiologicke centrum Multiscan, s.r.o., Pardubice
  - Fakultani Nemocnice Kralavske Vinohadry, Praque
- Hungary (4):
  - Allami Egeszseguegi Koezpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Radiologicke centrum Multiscan, Debrecen
  - Clinfan Ltd SMO, County Hospital Szekszard, Szekszárd
- Russia (5):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Blokhin Russian Oncology Research Center of Russian Academy of Medical Sciences, Moscow
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - Russian Research Centre of Radiology and Surgery, Saint Petersburg
  - Stavropol Territory Clinical Oncology Dispensary, Stavropol

REFERENCES:
- [Derived] Yardley DA, Ismail-Khan RR, Melichar B, Lichinitser M, Munster PN, Klein PM, Cruickshank S, Miller KD, Lee MJ, Trepel JB. Randomized phase II, double-blind, placebo-controlled study of exemestane with or without entinostat in postmenopausal women with locally recurrent or metastatic estrogen receptor-positive breast cancer progressing on treatment with a nonsteroidal aromatase inhibitor. J Clin Oncol. 2013 Jun 10;31(17):2128-35. doi: 10.1200/JCO.2012.43.7251. Epub 2013 May 6. PMID 23650416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 38 investigative sites in the United States, Canada, Czech Republic, Hungary and Russia from 13 June 2008 to 26 November 2012.
Pre-assignment Details: Participants with a diagnosis of metastatic breast cancer were enrolled equally in one of two treatment arms: exemestane 25 mg plus entinostat 5 mg or exemestane 25 mg plus placebo.
Period: Overall Study
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg
Started | 66 | 64
Completed | 21 | 26
Not Completed | 45 | 38
Not completed — Death | 43 | 27
Not completed — Withdrew Consent | 1 | 8
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.06) | 62.2 (11.72) | 62.4 (10.87)
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 2 | 3 | 5
  45 to 64 years | 38 | 32 | 70
  65 to 74 years | 19 | 19 | 38
  ≥75 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 65 | 61 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 5 | 4 | 9
  White | 61 | 60 | 121
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Height data is only available for n= 65, 63 participants.
  centimeters (cm)
    number analyzed (Participants) | 65 | 63 | 128
    (all) | 164.9 (6.38) | 162.7 (6.44) | 163.8 (6.48)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 73.2 (17.47) | 75.6 (16.66) | 74.3 (17.05)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance status is an assessment of a participant's general well-being and activities of daily of life. Scores range from 0=perfect health (asymptomatic; able to carry out activities without restriction) to 5=death.
  Participants
    Score=0 | 50 | 40 | 90
    Score=1 | 16 | 24 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the number of months from the date of randomization to the earlier of progressive disease (PD) or death due to any cause.
Time Frame: From date of randomization to discontinuation due to disease progression or death up to primary completion date (Median follow-up 6 months)
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg
Number analyzed (Participants) | 66 | 64
months | 2.27 [1.81 to 3.68] | 4.28 [3.26 to 5.36]
Statistical Analysis 1: Comparison: Exemestane 25 mg + Placebo vs Exemestane 25 mg + Entinostat 5 mg; Test type: Superiority; p = 0.06, Log Rank; P-value is stratified by the randomization stratification factors and is 1-sided, with a 0.10 threshold for significance; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.49 to 1.09]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with response during treatment classified as complete response (CR) or partial response (PR), as assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: From date of randomization to discontinuation due to disease progression or intolerable Adverse Event (AE) up to primary completion date (Median follow-up 6 months)
Population: Full Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg
Number analyzed (Participants) | 66 | 64
percentage of participants | 4.6 [1.0 to 12.7] | 4.7 [1.0 to 13.1]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as the percentage of participants with overall response (CR + PR) plus stable disease (SD) for 6 months as assessed by the investigator based on RECIST, version 1.0. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: From date of randomization to discontinuation due to disease progression or intolerable AE up to primary completion date (Median follow-up 6 months)
Population: Full Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg
Number analyzed (Participants) | 66 | 64
percentage of participants | 25.8 [15.8 to 38.0] | 26.6 [16.3 to 39.1]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Worsening of a pre-existing medical condition was considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. Abnormal clinical laboratory findings determined by the investigator to be clinically significant were recorded as AEs. A TEAE is an AE that starts after the administration of study drug.
  A SAE is any AE that is fatal, life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth effect or other significant medical hazard.
Time Frame: First dose to within 30 days of last dose of study drug (Up to Approximately 2 Years)
Population: Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg
Number analyzed (Participants) | 66 | 63
Participants
  TEAE | 56 | 60
  SAE | 8 | 10

5. Other Pre Specified Outcome: Overall Survival (OS)
Description: OS was defined as the number of months elapsed between the date of randomization and the date of death (whatever the cause).
Time Frame: First dose of study drug to end of study (Median follow-up 24 months in the EE arm and 26.4 months in the EP arm)
Population: Full Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Exemestane 25 mg + Placebo (EP): Exemestane (Aromasin®) 25 mg tablets orally once daily plus a placebo-matching entinostat tablet orally once per week on Days 1, 8, 15 and 22 of each 28-day treatment cycle until development of progressive disease (PD) or unacceptable toxicity or closure of the study by the Sponsor, whichever occurred first.
- Exemestane 25 mg + Entinostat 5 mg (EE): Exemestane (Aromasin®) 25 mg tablets orally once daily plus an entinostat 5 mg tablet orally once per week on Days 1, 8, 15 and 22 of each 28-day treatment cycle until development of progressive disease (PD) or unacceptable toxicity or closure of the study by the Sponsor, whichever occurred first.
Arm/Group | Exemestane 25 mg + Placebo (EP) | Exemestane 25 mg + Entinostat 5 mg (EE)
Number analyzed (Participants) | 66 | 64
months | 19.84 [17.04 to 26.71] | 28.13 [21.15 to NA] — Upper Confidence Interval was not estimable due to the low number of participants with events.
Statistical Analysis 1: Comparison: Exemestane 25 mg + Placebo (EP) vs Exemestane 25 mg + Entinostat 5 mg (EE); Test type: Superiority; p = 0.018, Log Rank — P-value is stratified by the randomization stratification factors and is 1-sided; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.36 to 0.97] — Hazard ratio was estimated from a Cox proportional hazards model. Placebo serves as the reference treatment group for the interpretation of the hazard ratio

ADVERSE EVENTS:
Time Frame: First dose to within 30 days of last dose of study drug (Up to approximately 2 Years)
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Exemestane 25 mg + Placebo | Exemestane 25 mg + Entinostat 5 mg
Serious Adverse Events (participants affected / at risk) | 8/66 | 10/63
Other Adverse Events (participants affected / at risk) | 51/66 | 58/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane 25 mg + Placebo (N=66) | Exemestane 25 mg + Entinostat 5 mg (N=63)
Anemia group (Blood and lymphatic system disorders) | 1 | 1
Lobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Leukopenia group (Blood and lymphatic system disorders) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Thrombocytopenia group (Blood and lymphatic system disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane 25 mg + Placebo (N=66) | Exemestane 25 mg + Entinostat 5 mg (N=63)
Anemia group (Blood and lymphatic system disorders) | 7 | 12
Neutropenia group (Blood and lymphatic system disorders) | 1 | 19
Thrombocytopenia group (Blood and lymphatic system disorders) | 3 | 12
Leukopenia group (Blood and lymphatic system disorders) | 1 | 9
Tachycardia (Cardiac disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 10 | 25
Diarrhoea (Gastrointestinal disorders) | 8 | 11
Constipation (Gastrointestinal disorders) | 10 | 6
Vomiting (Gastrointestinal disorders) | 3 | 13
Abdominal pain upper (Gastrointestinal disorders) | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 9
Fatigue (General disorders) | 17 | 30
Oedema peripheral (General disorders) | 3 | 13
Pain (General disorders) | 4 | 10
Hot flush (General disorders) | 6 | 5
Pyrexia (Gastrointestinal disorders) | 3 | 4
Asthenia (General disorders) | 4 | 3
Chills (General disorders) | 0 | 4
Weight decreased (Investigations) | 12 | 13
Blood alkaline phosphatase increased (Investigations) | 5 | 5
Aspartate aminotransferase increased (Investigations) | 7 | 3
Alanine aminotransferase increased (Investigations) | 6 | 3
Electrocardiogram QT prolonged (Investigations) | 6 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 5 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 7
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 7 | 9
Insomnia (Nervous system disorders) | 7 | 7
Neuropathy (Nervous system disorders) | 0 | 4
Anxiety (Psychiatric disorders) | 3 | 6
Urinary tract infection (Renal and urinary disorders) | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 4
Vascular disorders (Vascular disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the multi-center Study shall not be made before the first multi-site publication by Sponsor or Publications Committee. No Public Presentation by Institution or Investigator will be made until Study Documentation/Results from all sites are received and analyzed by Sponsor. Separate publication by Investigator will be delayed for a period of 18 months until the initial publication by Committee or Sponsor, or a determination is made not to make such publication.